CLINICAL TRIAL: NCT04392596
Title: Performance of Bone Mineral Density and Trabecular Bone Score in Assessment of Bone Quality in Egyptian Male Patients With Ankylosing Spondylitis
Brief Title: Study of Bone Mineral Density and Trabecular Bone Score in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 20201
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: AS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- patients (Experimental): 40
  Interventions: Device: Bone Mineral Density and Trabecular Bone score

INTERVENTIONS:
Device: Bone Mineral Density and Trabecular Bone score — structural damage in the cervical and lumbar spine was scored according to the modified Stoke AS Spinal Score (mSASSS) which yielded a final summation score ranging from zero to 72.
  BMD was measured using DXA (Lunar Prodigy densitometer, GE Healthcare, Madison, WI, USA).
  BMD was measured at the lumbar spine (L1-L4) and the left hip (femoral neck and total proximal femur).
  TBS was analyzed using DXA images over exactly the same region as the lumbar BMD assessment (L1-L4). Lumbar spine DXA images were reanalyzed using TBS iNight software version 2.1 (Med-I maps, Merignac, France). Patients were divided in 3 TBS groups according to guidelines for fracture risk [22]: any TBS >1.31 was considered as normal; TBS values between 1.23 and 1.31 were consistent as partially degraded structure; and any TBS <1.23 was considered as degraded structure.

SUMMARY:
Osteoporosis is a common complication of AS even in the early stages of disease. Yet, AS is also characterized by new bone growth that leads to syndesmophytes formation and subsequent vertebral ankyloses.

DETAILED DESCRIPTION:
Accordingly, previously-published studies have demonstrated large discrepancies in the reported incidence of osteoporosis, based on measurement of bone mineral density (BMD), in patients with AS ranging from 18.7% to 62%. Measurement of trabecular bone score (TBS) is a novel tool used to evaluate bone microarchitecture. Aim of the work: to compare bone quality using TBS between AS patients and healthy controls and to evaluate factors associated with TBS in patients with AS. Patients and methods: A total of 40 male AS patients recruited from Outpatient Clinic of Rheumatology, Mansoura University Hospital. 40 age-matched healthy males as matched control. TBS was analyzed using DXA images over exactly the same region as the lumbar BMD assessment (L1-L4). Lumbar spine DXA images were reanalyzed using TBS iNight software version 2.1 (Med-I maps, Merignac, France). Patients were divided in 3 TBS groups according to guidelines for fracture risk: any TBS >1.31 was considered as normal; TBS values between 1.23 and 1.31 were consistent as partially degraded structure; and any TBS <1.23 was considered as degraded structure

ELIGIBILITY:
Inclusion Criteria:

* A total of 40 consecutive male AS patients were invited to participate in this study. Patients were recruited from Outpatient Clinic of Rheumatology, Mansoura University Hospital, between January and September 2019. AS was diagnosed according to modified New York criteria. During the same period, 40 age-matched healthy males were invited to participate in the study as a control group.

Exclusion Criteria:

* patients or controls with thyroid or parathyroid disorders, presence of chronic renal or liver disease, and use of any medication that could potentially interfere with bone metabolism including bisphosphonates, teriparatide, anticonvulsants, anticoagulants, calcium and corticosteroids. None of the participants was using vitamin D supplements.

Ages: 22 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
to compare bone quality using TBS between AS patients and healthy controls and to evaluate factors associated with TBS in patients with AS | 1 year
  TBS was analyzed using DXA images over exactly the same region as the lumbar BMD assessment (L1-L4). Lumbar spine DXA images were reanalyzed using TBS iNight software version 2.1 (Med-I maps, Merignac, France). Patients were divided in 3 TBS groups according to guidelines for fracture risk: any TBS >1.31 was considered as normal; TBS values between 1.23 and 1.31 were consistent as partially degraded structure; and any TBS <1.23 was considered as degraded structure

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin AD Hussein, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data available upon request